CLINICAL TRIAL: NCT03309839
Title: HLA-DR Expression in Neonates After Cardiac Surgery Under Cardiopulmonary Bypass
Acronym: IMMUNOPED
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Fédération Française de Cardiologie (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0359
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Cardiac Surgery
Keywords: HLA-DR expression; cardiopulmonary bypass; neonate
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neonates with cardiac surgery under cardiopulmonary bypass
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — A sample of an additional blood tube will be taken in parallel with the blood test carried out for the treatment.

SUMMARY:
The purpose of this study is to determine how monocyte HLA-DR and other markers of immune function change with time in neonates who underwent cardiac surgery with cardiopulmonary bypasss.

We hypothesize that HLA-DR expression in neonates is predictive of septic complications after cardiopulmonary bypass

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≤ 28 days
* Admission after cardiac surgery under cardiopulmonary bypass

Exclusion Criteria:

* Lack of parental consent

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged ≤ 28 days after cardiac surgery under cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-04-13 (Actual)

PRIMARY OUTCOMES:
HLA-DR expression | Preoperatively, and 1, 2, 3 and 4 days after the end of cardiopulmonary bypass
  Number of HLA-DR molecules per monocyte (AB/c) determined by flow cytometry on whole blood using a Quantibrite phycoerythrin fluorescence quantitation kit (BD Biosciences) Number of HLA-DR molecules per monocyte (AB/c) determined by flow cytometry on whole blood using a Quantibrite phycoerythrin fluorescence quantitation kit (BD Biosciences)

SECONDARY OUTCOMES:
Cytokines measurements | Preoperatively, and 1, 2, 3 and 4 days after the end of cardiopulmonary bypass
  Pro and anti-inflammatory cytokine concentrations in the plasma measured by multiplex immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Chenouard, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No